CLINICAL TRIAL: NCT04384432
Title: Effectiveness of Routine Physical Therapy With and Without Thoracic Mobility Exercises in Patients With Chronic Neck Pain
Brief Title: Effectiveness of Routine Physical Therapy With and Without Thoracic Mobility Exercises in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Ishtiaq Ahmed, Physiotherapist, Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 247
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Neck Pain
Keywords: THORACIC MOBILITY EXERCISES; Chronic Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Physical Therapy with Thoracic mobility exercise (Experimental): Combination of Routine Physical Therapy with Thoracic mobility exercise.
  Interventions: Other: Routine Physical Therapy with Thoracic mobility exercise
- Routine Physical Therapy (Active Comparator): Routine Physical Therapy exercise
  Interventions: Other: Routıne Physıcal therapy

INTERVENTIONS:
Other: Routine Physical Therapy with Thoracic mobility exercise — Combınatıon of routıne Routine Physical Therapy with Thoracic mobility exercise
  Arms: Routine Physical Therapy with Thoracic mobility exercise
Other: Routıne Physıcal therapy — Exercise for Chronic Neck Pain
  Arms: Routine Physical Therapy

SUMMARY:
There is a limited data available on the effectiveness of thoracic mobility exercises in chronic neck pain and there is a need to determine these exercises in chronic neck pain because chronic neck pain has significant effects on the surrounding muscles of the neck and cervical spine and along with the muscles of shoulder and arm. So the mobility exercises of any region around the neck area can reduce neck pain because these structures are interlinked anatomically and functionally aspects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* A medical diagnosis of chronic cervical pain (more than 3 months of cervical pain evolution)
* Positive flexion rotation test

Exclusion Criteria:

* cervical radiculopathy
* History of Trauma, any Surgery, any Systemic diseases, any Fractures, congenital diseases.
* Dislocation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Neck Disability Index Questionnaire | 8 week
  The Neck Disability Index is a modification of the Oswestry Low Back Pain Disability Index . It is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. The Neck Disability Index has sufficient support and usefulness to retain its current status as the most commonly used self-report measure for neck painç maximum Score is 50.
  0 - 4 = no disability 5 - 14 = mild 15 - 24 = moderate 25 - 34 = severe above 34 = complete.
Visual Analogue Scale | 8 week
  To determine the change in pain of patients. Total score is 10. Higher the score, Greater the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Awais Bin Inam, MSOMPT, Study Director — Government College University
Locations (1):
- Suraiya Majeed Trust hospital and Bin Inam clinic, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No